CLINICAL TRIAL: NCT04241601
Title: Low-dose Interleukin-2 for the Reduction of Vascular Inflammation in Acute Coronary Syndromes
Brief Title: Low-dose Interleukin-2 for the Reduction of Vascular Inflammation in Acute Coronary Syndromes - IVORY
Acronym: IVORY
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Cambridge University Hospitals NHS Foundation Trust (Other)
Responsible Party: Principal Investigator, Joseph Cheriyan, MBChB, MA, FRCP, FESC, FACC, Consultant Physician & Clinical Pharmacologist/Affiliated Assoc Professor, Cambridge University Hospitals NHS Foundation Trust
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IVORY; 2017-005130-27 (EudraCT Number)
Record Dates: First submitted 2019-12-09; First posted 2020-01-27 (Actual); Last update posted 2024-06-10 (Actual); Status verified 2024-06

CONDITIONS: Acute Coronary Syndromes
Keywords: Acute Coronary Syndromes
MeSH Terms: conditions — Acute Coronary Syndrome | interventions — Interleukin-2; aldesleukin; Solutions

STUDY DESIGN:
Intervention Model Description: a randomised, double-blind, placebo controlled, parallel group experimental medicine trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The trial will be double-blind, with active and placebo doses appearing identical at point of issue and administration. The CUH central pharmacy will be unblinded and provided with a copy of the concealment list. Data analysis for the trial will be performed by a statistician who will be unblinded after the database lock.
  The statistician, or delegate, may be unblinded for individual patients after their treatment period has concluded, to facilitate rapid reporting of safety events.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- low dose interleukin-2 (Active Comparator): Commercially available aldesleukin with a UK marketing authorisation will be used and will be initially prepared as per SmPC. Active and Placebo doses appearing identical at point of issue and administration.
  Interventions: Drug: Interleukin-2 [IL-2]
- Placebo (Placebo Comparator): Commercially available dextrose 5% injection with a UK marketing authorisation at equivalent dose volume will be used for the placebo formulation. Placebo and Active doses appearing identical at point of issue and administration.
  Interventions: Other: Placebo Dextrose 5% solution

INTERVENTIONS:
Drug: Interleukin-2 [IL-2] — Active Comparator: IL-2 plays a key role in Treg cell development, expansion, survival and suppressive function
  Other Names: Aldesleukin
  Arms: low dose interleukin-2
Other: Placebo Dextrose 5% solution — Placebo Comparator: Dextrose 5% solution
  Arms: Placebo

SUMMARY:
Acute coronary syndromes (ACS) result from coronary plaque(s) disruption, which initiates a thrombotic process leading to partial or complete obstruction of the vessel lumen with subsequent myocardial ischaemia and necrosis. The mainstay of treatment is currently focused on the re-establishment and maintenance of coronary artery patency using anti-platelets and anticoagulants with or without mechanical dilatation and stenting of the culprit artery. Despite important advances in management, ACS still carries a risk of substantial morbidity and mortality. The improved efficacy of novel anti-platelet and anticoagulant agents have been limited by increased risk of haemorrhagic events. Future breakthroughs in management are most likely to arise from targeting other relevant pathophysiological pathways. Particularly, the immune response which is an important process that has been neglected in the management of patients with ACS.

In this trial the investigators investigate the efficacy of low dose IL-2 compared with placebo in patients with ACS.

DETAILED DESCRIPTION:
A heart attack occurs when there is reduced blood flow to heart muscle cells which results from narrowings or blockages in walls of blood vessels supplying the heart, due to fatty deposits and inflammatory cells that build up over time. This build-up leads to heart muscle damage called a heart attack. The immune system plays an important role in both the development of the narrowings and the damage to the heart muscle during a heart attack. Studies have shown that there is a lower level of protective immune cells called regulatory T-cells (Tregs) in heart attack patients. Increasing the number of circulating Tregs may have a direct effect in reducing the inflammation in arteries, preventing further narrowings in blood vessels and improving heart muscle function.

Aldesleukin, also known as interleukin-2 (IL-2), is a medicine that stimulates the production of Treg cells when given at low doses and is the drug being tested in this trial. IL-2 is licensed for the treatment of kidney cancer where it is given at much higher doses than planned in this trial. It appears to be safe and well tolerated at low doses while increasing Treg cells.

IVORY will be conducted in patients presenting with a heart attack (Acute Coronary Syndrome (ACS)). Approximately, 60 patients will be randomized to receive either low dose IL-2 or placebo. It is a Phase 2, randomised, double- blinded, placebo-controlled experimental trial. Total study duration for each participant will be approximately 13 weeks.

Participants will undergo two PET/CT (Positron emission tomography-computed tomography) scans to observe change of inflammation in the blood vessels from baseline between the two trial groups (Primary Endpoint).

ELIGIBILITY:
Inclusion Criteria:

* Able to provide written informed consent to participate.
* Current admission (on the screening visit) with an acute coronary syndrome - ST elevation myocardial infarction (STEMI), non-ST elevation myocardial infarction (NSTEMI), or unstable angina (UA) with symptoms suggestive of myocardial ischaemia lasting 10 minutes or longer with the patient at rest or with minimal effort AND EITHER i. elevated levels of TnI on admission OR ii. dynamic changes in ECG (new ST-T changes or T-wave inversion).
* Where applicable, to be included in the trial women must be:

  i) Postmenopausal (for the purposes of this trial, postmenopausal is defined as being amenorrhoeic for greater than 2 years with an appropriate clinical profile, e.g. age appropriate, history of vasomotor symptoms) OR ii) Have had a documented hysterectomy and/or bilateral oophorectomy or sterilised OR iii) Peri-menopausal with a negative pregnancy test at screening (for the purposes of inclusion in this trial. Peri-menopausal is defined as women with an appropriate clinical profile, e.g. age appropriate, history of vasomotor symptoms, irregular periods). They will also have to comply with the use of contraception for the duration of the trial and undergo additional pregnancy tests during and after treatment.
* High sensitivity C-reactive protein of >2 mg/L at any point from index admission for acute event to screening (inclusive).
* Willingness and possibility to start dosing within 14 days from initial date of admission to the primary hospital for ACS.
* Able to comply with all trial mandated visits.

Exclusion Criteria:

* Current presentation (at screening) with cardiogenic shock (systolic blood pressure <80 mm Hg, unresponsive to fluids, or necessitating catecholamines).
* Current presentation with cardiac arrest.
* Signs or symptoms of active infection requiring intravenous antibiotic treatment at screening.
* History of malignancies requiring active treatment (However, patients with a history of treated localised basal or squamous cell skin cancer are not excluded from participation in this trial).
* History of solid organ transplantation or other bone marrow transplantation.
* History of recurrent epileptic seizures in the previous 4 years; repetitive or difficult to control seizures, coma or toxic psychosis lasting >48 hours.
* Uncontrolled hypotension (Systolic BP (SBP)<80mmHg or DBP<50mmHg) OR uncontrolled hypertension (SBP>180 or DBP>120 mmHg) at screening.
* Average corrected QT interval (QTc) > 450 msecs using Bazett's formula from average of triplicate ECGs (or > 480 msecs if bundle branch block).
* Renal impairment defined as Creatinine clearance [Cockcroft-Gault] <45ml/min at screening.
* Liver dysfunction (defined as ALT > 2xULN) at screening.
* Evidence of cholestasis defined as elevated Total Bilirubin Levels, (TBL > 1.5 x ULN) and Alkaline Phosphatase, ALP (ALP > 1.5 x ULN), at screening.
* Known hypothyroidism or hyperthyroidism.
* Known autoimmune disease requiring active immunosuppressive treatment.
* Any oral or intravenous immunosuppressive treatment including regular prednisolone, hydrocortisone or disease modifying drugs. [Inhaled or topical steroids are permissible].
* Patients on cytotoxic drugs and interferon-alpha.
* Diabetics on oral hypglycaemics/diet control with HbA1c (DCCT) >8% (OR HbA1c (IFCC) >64mmol/mol) at screening. Diabetics on insulin are excluded from the study.
* Contraindication to IL-2 treatment or hypersensitivity to IL-2 or to any of its excipients.
* Participation in a previous research trial in the last 3 years which involved exposure to significant ionising radiation (i.e. cumulative research radiation dose >5 mSv)
* Participation in a clinical trial where the patient has received a drug or new chemical entity within 30 days or 5 half-lives, or twice the duration of the biological effect of the drug (whichever is longer) prior to the first dose of trial medication, Visit 3 (Day 1).
* Any medical history or clinically relevant abnormality that is deemed by the principal investigator/delegate to make the patient ineligible for inclusion because of a safety concern.
* Pregnant women or breast feeding women.
* Patients who are COVID-19 PCR positive at the time of screening.
* Known severe allergy to the CT-contrast agents.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2020-08-05 (Actual); Primary Completion 2023-01-25 (Actual); Study Completion 2023-01-25 (Actual)

PRIMARY OUTCOMES:
Change in vascular inflammation | Baseline: Visit 2, day -6-0, and Follow Up: Visit 15, day 61
  Vascular inflammation (as measured by mean TBR max in the index vessel) is measured by mean TBR max in the index vessel by 18F-FDG PET/CT

SECONDARY OUTCOMES:
Change in mean TBR max in each arterial region | Baseline: Visit 2, day -6-0, and Follow Up: Visit 15, day 61
  Change in mean max TBR in each arterial region individually restricted to those slices with TBR>1.6
Change in lymphocyte subsets | Throughout treatment period: Visit 3, day 1; Visit 7, day 5; Visit 8, day 12; Visit 10, day 26; Visit 12, day 40; Visit 14, day 54, Visit 15, day 61
  Lymphocyte subsets:T effector [Teffs] cells defined as central memory and effector memory T cells in the non-Treg gated T cells. Evaluated by flow cytometry
Change in percentage of Treg cells between low dose IL-2 and placebo | Throughout treatment period: Visit 3, day 1; Visit 7, day 5; Visit 8, day 12; Visit 10, day 26; Visit 12, day 40; Visit 14, day 54, Visit 15, day 61.
  Treg cells are defined as CD3+CD4+CD25highCD127low cells within the CD3+CD4+ T cell gate. Evaluated by flow cytometry
Extended dosing of IL-2 in ACS patients safety and tolerability: Incidence of Adverse Events | Visit 1 (day -14-0) through to Visit 16 (day 82)
  Number of incidences of adverse events is assessed via adverse change in routine test results and patient consultation. Events will be catalogued using MedDRA coding.
Extended dosing of IL-2 in ACS patients safety and tolerability: Incidence of injection site reaction | All dosing visit: Visit 3 (day 1) through to Visit 14 (day 54)
  Location of injection site will be recorded as will incidences of induration, redness and swelling at the injection site
Extended dosing of IL-2 in ACS patients safety and tolerability: Full Blood Count: total white cell count | Baseline, Visit 3 (day 1) thorugh Visit 14 (day 54) and Visit 16 (day 82 when clinically indicated and patient attends hospital)
  Haematology tests - full blood count: Total white cell count (WBC), in 10^9/L
Extended dosing of IL-2 in ACS patients safety and tolerability: Full Blood Count: Red cell count | Baseline, Visit 3 (day 1) thorugh Visit 14 (day 54) and Visit 16 (day 82 when clinically indicated and patient attends hospital)
  Haematology tests - full blood count: Red cell count (RBC), in 10^12/L
Extended dosing of IL-2 in ACS patients safety and tolerability: Full Blood Count: Haemoglobin | Baseline, Visit 3 (day 1) thorugh Visit 14 (day 54) and Visit 16 (day 82 when clinically indicated and patient attends hospital)
  Haematology tests - full blood count: Haemoglobin (Hb), in g/L
Extended dosing of IL-2 in ACS patients safety and tolerability: Full Blood Count: Platelets | Baseline, Visit 3 (day 1) thorugh Visit 14 (day 54) and Visit 16 (day 82 when clinically indicated and patient attends hospital)
  Haematology tests - full blood count: Platelet Count, in 10^9/L
Extended dosing of IL-2 in ACS patients safety and tolerability: Differential blood count - Neutrophils | Baseline, Visit 3 (day 1) thorugh Visit 14 (day 54) and Visit 16 (day 82 when clinically indicated and patient attends hospital)
  Haematology tests - differential blood count: Neutrophils, in 10^9/L
Extended dosing of IL-2 in ACS patients safety and tolerability: Differential blood count - Lymphocytes | Baseline, Visit 3 (day 1) thorugh Visit 14 (day 54) and Visit 16 (day 82 when clinically indicated and patient attends hospital)
  Haematology tests - differential blood count: Lymphocytes, in 10^9/L
Extended dosing of IL-2 in ACS patients safety and tolerability: Differential blood count - Monocytes | Baseline, Visit 3 (day 1) thorugh Visit 14 (day 54) and Visit 16 (day 82 when clinically indicated and patient attends hospital)
  Haematology tests - differential blood count: Monocytes, in 10^9/L
Extended dosing of IL-2 in ACS patients safety and tolerability: Differential blood count - Eosinophils | Baseline, Visit 3 (day 1) thorugh Visit 14 (day 54) and Visit 16 (day 82 when clinically indicated and patient attends hospital)
  Haematology tests - differential blood count: Eosinophils, in 10^9/L
Extended dosing of IL-2 in ACS patients safety and tolerability: Differential blood count - Basophils | Baseline, Visit 3 (day 1) thorugh Visit 14 (day 54) and Visit 16 (day 82 when clinically indicated and patient attends hospital)
  Haematology tests - differential blood count: Basophils, in 10^9/L
Extended dosing of IL-2 in ACS patients safety and tolerability: Clinical biochemistry - Urea | Baseline, Visit 3 (day 1) through Visit 14 (day 54) and Visit 16 (day 82 when clinically indicated and patient attends hospital)
  Clinical biochemistry test: level of urea, in mmol/L
Extended dosing of IL-2 in ACS patients safety and tolerability: Clinical biochemistry - Creatinine | Baseline, Visit 3 (day 1) through Visit 14 (day 54) and Visit 16 (day 82 when clinically indicated and patient attends hospital)
  Clinical biochemistry test: level of creatinine, in µmol/L
Extended dosing of IL-2 in ACS patients safety and tolerability: Clinical biochemistry test for liver function - ALT | Baseline, Visit 3 (day 1) through Visit 14 (day 54) and Visit 16 (day 82 when clinically indicated and patient attends hospital)
  Clinical biochemistry blood test for liver function: Alanine Aminotransferase (ALT), in µ/L
Extended dosing of IL-2 in ACS patients safety and tolerability: Clinical biochemistry test for liver function - ALP | Baseline, Visit 3 (day 1) through Visit 14 (day 54) and Visit 16 (day 82 when clinically indicated and patient attends hospital)
  Clinical biochemistry blood test for liver function: Alkaline Phosphatase (ALP), in µ/L
Extended dosing of IL-2 in ACS patients safety and tolerability: Clinical biochemistry test for liver function - Albumin | Baseline, Visit 3 (day 1) through Visit 14 (day 54) and Visit 16 (day 82 when clinically indicated and patient attends hospital)
  Clinical biochemistry blood test for liver function: Albumin, in g/L
Extended dosing of IL-2 in ACS patients safety and tolerability: Clinical biochemistry test for liver function - Bilirubin | Baseline, Visit 3 (day 1) through Visit 14 (day 54) and Visit 16 (day 82 when clinically indicated and patient attends hospital)
  Clinical biochemistry blood test for liver function: Bilirubin, in µmol/L
Extended dosing of IL-2 in ACS patients safety and tolerability: Thyroid function | Visit 1 (day -14-0)
  A thyroid function blood test of level of TSH (thyroid-stimulating hormone) in the blood will be performed. T4 (Thyroxine) will be performed if TSH is abnormal.
Extended dosing of IL-2 in ACS patients safety and tolerability: Electrical activity of the heart recorded using a 12-lead electrocardiogram | Baseline, Visit 3 (day 1) through Visit 14 (day 54), and Visit 16 (day 82 when clinically indicated and patient attends hospital)
  12-lead ECG recording - QTcB (Corrected QT using Bazett's formula) intervals, in ms
Extended dosing of IL-2 in ACS patients safety and tolerability: Blood pressure assessment | Baseline, Visit 3 (day 1) through Visit 14 (day 54), and Visit 16 (day 82 when clinically indicated and patient attends hospital)
  Blood pressure will be assessed using systolic and diastolic pressure measured in mmHg.
Extended dosing of IL-2 in ACS patients safety and tolerability: Heart rate assessment | Baseline, Visit 3 (day 1) through Visit 14 (day 54), and Visit 16 (day 82 when clinically indicated and patient attends hospital)
  Heart rate assessed using bpm
Extended dosing of IL-2 in ACS patients safety and tolerability: Respiratory rate assessment | Baseline, Visit 3 (day 1) through Visit 14 (day 54), and Visit 16 (day 82 when clinically indicated and patient attends hospital)
  Measured using breaths per minute
Extended dosing of IL-2 in ACS patients safety and tolerability: Oxygen saturation assessment | Baseline, Visit 3 (day 1) through Visit 14 (day 54), and Visit 16 (day 82 when clinically indicated and patient attends hospital)
  Assessment of oxygen saturation and measured in percentage
Extended dosing of IL-2 in ACS patients safety and tolerability: Physical examination evaluation - Gastrointestinal | Baseline, Visit 3 (day 1) through Visit 14 (day 54), and Visit 16 (day 82 when clinically indicated and patient attends hospital)
  Incidences of a abdominal distention, palpations and/or patient self-report of physical discomfort or pain
Extended dosing of IL-2 in ACS patients safety and tolerability: Physical examination evaluation - Skin | Baseline, Visit 3 (day 1) through Visit 14 (day 54), and Visit 16 (day 82 when clinically indicated and patient attends hospital)
  Incidences of ISR lesions, nodules and/or bruising
Extended dosing of IL-2 in ACS patients safety and tolerability: Incidence of cardiovascular events | Visit 2 (day -6-0) and Visit 15 (day 61)
  Occurrence of another important cardiovascular event(s) such a myocardial infarction. These will be captured through AEs and SAEs

OTHER OUTCOMES:
Change in serum cardiac biomarkers: hsCRP | Throughout treatment period: Visit 3, day 1; Visit 7, day 5; Visit 8, day 12; Visit 10, day 26; Visit 12, day 40; Visit 14, day 54; Visit 15, day 61.
  High-sensitivity C-reactive protein (hsCRP), in mg/L
Change in serum cardiac biomarkers: IL-6 | Throughout treatment period: Visit 3, day 1; Visit 7, day 5; Visit 8, day 12; Visit 10, day 26; Visit 12, day 40; Visit 14, day 54; Visit 15, day 61.
  Interleukin 6 (IL-6), in pg/ml
Change in serum cardiac biomarkers: Troponin I | Throughout treatment period: Visit 3, day 1; Visit 7, day 5; Visit 8, day 12; Visit 10, day 26; Visit 12, day 40; Visit 14, day 54; Visit 15, day 61.
  Troponin I, in ng/L
Change in ejection fraction | Visit1 day -14 to day 0; visit 14 (can be done between visit 14 and 16)
  Change in ejection fraction. Measures on transthoracic echocardiograms
Change in phenotype and function of peripheral blood mononuclear cell subsets | Throughout treatment period: Visit 3, day 1; Visit 7, day 5; Visit 8, day 12; Visit 10, day 26; Visit 12, day 40; Visit 14, day 54; Visit 15, day 61.
  Change in phenotype and function of peripheral blood mononuclear cell (PBMC) subsets (such as B lymphocytes and Natural Killer cells). Assessed by flow cytometry, gene expression, in vitro activation and suppression assays
Differences in gut microbiota composition between low-dose IL-2 vs placebo | Visit 3, day 1 and Visit 15, day 61
  Differences in gut microbiota composition between low-dose IL-2 vs placebo will be identified using 16S- RNAseq. Assessed by stool sample.
The effect of low-dose IL-2 on coronary artery inflammation | Visit 15, day 61
  The effect of low-dose IL-2 on coronary artery inflammation, measured by perivascular fat attenuation using computed tomography coronary angiography.
The effect of low-dose IL-2 on 18F-FDG uptake in cervical/thoracic vertebrae | Visit 2, day -6-0 and Visit 15, day 61
  The effect of low-dose IL-2 on 18F-FDG uptake in cervical/thoracic vertebrae. Assessed by FDG PET/CT scan.

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Cheriyan, MBChB,FRCP, Principal Investigator — Cambridge Unversity Hospitals NHS Foundation Trust; Unversity of Cambridge
Locations (1):
- Addenbrooke's Hospital, Cambridge, Cambridgeshire, United Kingdom

REFERENCES:
- [Derived] Sriranjan-Rothwell RS, Zhao TX, Hoole SP, Bond SJ, Tarkin JM, Brubert J, Hubsch A, Helmy J, Bumanlag-Amis E, Jalaludeen N, Templin H, Jiang W, Tedgui A, Zhao X, Nus M, Warnes V, Krishnan U, O'Brien JW, Wall C, Rudd JHF, Cheriyan J, Mallat Z; IVORY investigators. Anti-inflammatory therapy with low-dose IL-2 in acute coronary syndromes: a randomized phase 2 trial. Nat Med. 2026 Jan 8. doi: 10.1038/s41591-025-04090-y. Online ahead of print. PMID 41507574
- [Derived] Tsiantoulas D, Binder CJ. Identifying the sensor elements of regulatory T cells in atherosclerosis. Nat Cardiovasc Res. 2024 Feb;3(2):106-107. doi: 10.1038/s44161-023-00416-6. No abstract available. PMID 39196191
- [Derived] Sriranjan R, Zhao TX, Tarkin J, Hubsch A, Helmy J, Vamvaka E, Jalaludeen N, Bond S, Hoole SP, Knott P, Buckenham S, Warnes V, Bird N, Cheow H, Templin H, Cacciottolo P, Rudd JHF, Mallat Z, Cheriyan J. Low-dose interleukin 2 for the reduction of vascular inflammation in acute coronary syndromes (IVORY): protocol and study rationale for a randomised, double-blind, placebo-controlled, phase II clinical trial. BMJ Open. 2022 Oct 7;12(10):e062602. doi: 10.1136/bmjopen-2022-062602. PMID 36207050